CLINICAL TRIAL: NCT05651789
Title: Randomized Controlled Trial on the Effectiveness and Safety of Carvedilol vs. Propranolol Combined With Endoscopic Treatment in Second Prophylaxis of Variceal Bleeding in Cirrhosis
Brief Title: Carvedilol vs. Propranolol in Second Prophylaxis of Variceal Bleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Collaborators: Chengdu Shangjin Nanfu Hospital (Unknown); West China Tianfu Hospital (Unknown)
Responsible Party: Principal Investigator, luo xuefeng, Professor of Hepatology, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NSBB-RVB
Record Dates: First submitted 2022-11-21; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Portal Hypertension; Varice Bleed; Cirrhosis, Liver
MeSH Terms: conditions — Hypertension, Portal; Liver Cirrhosis | interventions — Carvedilol; Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carvedilol (Experimental): Carvedilol is started at a dose of 6.25mg/d, and titrated to a maximum dose of 12.5mg/d. Doses are increased 3 days later. Avoid systolic blood pressure <90 mmHg.
  Interventions: Drug: Carvedilol
- Propranolol (Active Comparator): Propranolol is started at a dose of 20 mg/d and the dose will be increased by 10 mg twice a day steps every 2-3 days until the target (heart rate: 55~60 bpm) or to a maximum dose of 160 mg/d. Systolic arterial pressure is not less than 90 mm Hg and heart rate is not less than 50 bpm.
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Carvedilol — Carvedilol is started at a dose of 6.25mg/d, and titrated to a maximum dose of 12.5mg/d. Doses are increased 3 days later. Avoid systolic blood pressure <90 mmHg.
  Other Names: carvedilol as the nonselective beta-blockers
  Arms: Carvedilol
Drug: Propranolol — Propranolol is started at a dose of 20 mg/d and the dose will be increased by 10 mg twice a day steps every 2-3 days until the target (heart rate: 55~60 bpm) or to a maximum dose of 160 mg/d. Systolic arterial pressure is not less than 90 mm Hg and heart rate is not less than 50 bpm.
  Other Names: propranolol as the nonselective beta-blockers
  Arms: Propranolol

SUMMARY:
This randomized controlled trial was conducted to evaluate the efficacy and safety of carvedilol versus propranolol, combined with routine endoscopic treatment, in the secondary prophylaxis of variceal bleeding in patients with cirrhosis.

DETAILED DESCRIPTION:
Non-selective beta blockers combined with endoscopic variceal band ligation (EVL) is the most effective methods for the prevention of variceal bleeding. Carvedilol has emerged as the preferred NSBB for treating portal hypertension in compensated cirrhosis due to strong evidence demonstrating that it has a more pronounced effect than propranolol to reduce the hepatic vein pressure gradient (HVPG), together with good patient acceptability and safety profile. However, No data from prospectively designed trials are available on the efficacy of carvedilol in the secondary prophylaxis of variceal bleeding. The aim of this randomized controlled trial was to evaluate the effectiveness and safety of carvedilol compared to propranolol as secondary prophylaxis of variceal bleeding in patients with cirrhosis. All cirrhotic patients with at least one episode of variceal bleeding were included and randomized to the carvedilol or propranolol groups. EVL protocol was routinely performed in both groups. Variceal rebleeding, further decompensation, liver-related death, and overall survival was the outcomes of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 80 years old;
* With liver cirrhosis diagnosed by previous biopsy or by clinical criteria, and analytical image;
* At least 5 days after index variceal bleeding;
* Informed consent.

Exclusion Criteria:

* Refusal to participate in the study;
* Portal hypertension resulting from other causes than liver cirrhosis;
* More than 42 days after index variceal bleeding;
* Bleeding from cardiofundal gastric varices;
* Portal venous thrombosis >50% of the portal vein trunk;
* Contraindications to beta-blockers (asthma, chronic obstructive pulmonary disease, atrioventricular block, heart failure, bradycardia with HR ≤40 bpm, arteria hypotension with systolic blood pressure <90 mm Hg, peripheral arterial disease, uncontrolled diabetes);
* Prior NSBB+EVL combined treatment, TIPS implantation or surgical shunt as secondary prophylaxis of variceal bledding;
* Chronic kidney disease;
* Pregnancy or lactation;
* Neoplastic disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Variceal rebleeding rate | 1 year
  Acute variceal rebleeding rate at 1 year

SECONDARY OUTCOMES:
Further decompensation rate | 1 year
  This is a composite outcome that refers to rate of all further liver decompensation events at 1 year, including variceal rebleeding, recurrent or developement of ascites (grade≥2), overt hepatic encephalopathy, spontaneous bacterial peritonitis, acute kidney injury, acute-on-chronic liver failure, and liver-related death.
Adverse events | 1 year
  Hypotension (systolic blood pressure <90 mmHg or mean arterial pressure <65 mmHg), development of acute kidney injury/ hepatorenal syndrome, hyponatremia, weakness, shortness of breath, dizziness, gastrointestinal symptoms (nausea, constipation), or sexual and erectile dysfunction.
Transplant-free survival rate | 1 year
  The transplant-free survival rate at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xuefeng Luo, M.D., Principal Investigator — West China Hospital

IPD SHARING:
Plan to Share IPD: No